CLINICAL TRIAL: NCT06127147
Title: Effects of High-intensity Inspiratory Muscle Training as a Pre-cardiac Rehabilitation Intervention on Cardiovascular Functions in Patients With Heart Disease
Brief Title: High-intensity Inspiratory Muscle Training as a Pre-cardiac Rehabilitation in Heart Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: The Scientific and Technological Research Council of Turkey (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY2023-1089
Record Dates: First submitted 2023-11-06; First posted 2023-11-13 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Bypass Graft; CABG
Keywords: coronary artery bypass graft; inspiratory muscle training; endothelial function; arterial stiffness; CABG

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Study Group (Experimental): Patients who will perform inspiratory muscle training (IMT) with %60 of MIP intensity
  Interventions: Device: IMT
- Sham Group (Sham Comparator): Patients who will perform Sham-IMT
  Interventions: Device: Sham-IMT

INTERVENTIONS:
Device: IMT — The IMT protocol will consist of high-intensity daily training - 2 sets of 30 breaths with a 1-minute rest between sets, twice a day for 4 weeks using an IMT Threshold device (Threshold IMT Philips® Respironics, Inc). The intensity of the training will be set to 60% of each patient's maximal inspiratory pressure.
  Arms: Study Group
Device: Sham-IMT — The sham IMT protocol will consist of high-intensity daily training - 2 sets of 30 breaths with a 1-minute rest between sets, twice a day for 4 weeks using an IMT Threshold device (Threshold IMT Philips® Respironics, Inc) without intensity.
  Arms: Sham Group

SUMMARY:
Background/aim: Endothelial function is closely associated with coronary artery health among individuals being treated for heart disease. An impairment in endothelial function promotes arterial stiffening that directly contributes to elevated systolic blood pressure as a result of increased vascular resistance. Inspiratory muscle training is simply a form of training consisting of repeated inspirations against resistance. Inspiratory muscle training has also been applied to patients with chronic disease or as an additional therapy for cardiac rehabilitation and it has proven to be safe in these groups. Few studies in the literature examined the effects of high-intensity inspiratory muscle training in this population, however, these studies did not examine the direct effects of inspiratory muscle training on vascular function. To the best of our knowledge, the effects of inspiratory muscle training in patients with heart disease on endothelial function and arterial stiffness prior to starting cardiac rehabilitation have not been investigated. This study aims to investigate and interpret whether high-intensity inspiratory muscle training, beyond the usual care of heart disease, improves endothelial function and arterial stiffness.

Methods: The study was designed as a randomized controlled trial. Patients will be allocated for inspiratory muscle training (IMT) with 60% of maximum inspiratory pressure (MIP) or sham inspiratory muscle training (Sham-control), for 4 weeks. In both groups, before and after 4-week training, cardiovascular functions will be measured and compared.

DETAILED DESCRIPTION:
Background: Cardiovascular diseases (CVD) remain a leading cause of morbidity and mortality in both men and women in developed and developing societies (Joseph et al., 2017). Some degree of pulmonary dysfunction is highly likely in patients with heart disease compared to those without(Calles et al., 2016; Cahalin and Arena, 2015). This can affect pulmonary function, and gas exchange, as well as decrease maximum inspiratory and expiratory pressures (MIP and MEP, respectively)(Dos Santos et al., 2019; Haeffener et al., 2008; Roncada et al., 2015; Cahalin and Arena, 2015).

Inspiratory muscle training has been shown to be an effective form of training that enhances lung function. It consists of repetitive breath cycles where one inspires against resistance placed by a device and expires against no resistance. Studies that have applied this form of training in patients with heart disease have found significant improvements in MIP-MEP, tidal volume, vital capacity, and 6-minute walking distance. Few studies have examined the effects of high-intensity (between 50-80% of MIP) inspiratory muscle training in patients with heart disease (Dos Santos et al., 2019; Dos Santos et al., 2021; Laoutaris et al., 2007; Miozzo et al., 2018; Sadek et al., 2022). This level of training has been associated with greater improvements in the aferomentioned outcomes of interest, however, no study has explored the effects of high-intensity inspiratory muscle training in patients with heart disease on measures of cardiovascular function.

Aim: This study aims to investigate and interpret whether high-intensity inspiratory muscle training, beyond the usual care, improves endothelial function and arterial stiffness on cardiovascular function in patients with heart disease.

Methods: The study was designed as a randomized controlled trial. After coronary artery bypass graft surgery, patients will be invited to the study. The demographic and clinical characteristics of the patients will be recorded after consent is obtained from the volunteer patients who meet the inclusion criteria. Subsequently, patients will be randomly divided into two groups for inspiratory muscle training (IMT) with 60% maximum inspiratory pressure (MIP) or sham inspiratory muscle training (Sham-control), for 4 weeks. In both groups, before and after 4-week training, resting blood pressure (systolic/diastolic), resting heart rate, endothelial function, arterial stiffness, functional exercise capacity, the severity of dyspnea, and inspiratory muscle functions will be measured.

ELIGIBILITY:
Inclusion Criteria:

* Aged >18 years old
* Be able to walk independently.
* Had coronary artery bypass graft (CABG) surgery, history of percutaneous coronary interventions, heart failure, and/or myocardial infarction.
* Sufficient English language comprehension and cognitive ability to understand the study protocol, give informed consent and follow instructions.

Exclusion Criteria:

* Being a current smoker (or tobacco).
* Having a diagnosed chronic disease such as inflammatory bowel disease/irritable bowel syndrome, cerebrovascular diseases, COPD, chronic kidney disease requiring dialysis, neurological disorders, or diseases that may affect motor/cognitive function [multiple sclerosis, Parkinson's disease, polio, Alzheimer's disease, dementia, or other brain diseases of ageing])
* Getting a score below 24 on the Standardized Mini Mental Test
* Using antipsychotic medications commonly used to treat schizophrenia or schizoaffective disorders (i.e., haloperidol)
* Having had any other previous cardiothoracic operation except CABG (e.g. Pneumonectomy, lobectomy, etc.)
* Having a history of unstable-angina
* Having had pneumonia in the last 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-06-07 (Actual); Study Completion 2024-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cemal Ozemek, Assoc. Prof., Principal Investigator — University of Illinois at Chicago
Locations (2):
- United States (2):
  - University of Illinois at Chicago, Chicago, Illinois
  - University of Illinois Chicago, Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dos Santos TD, Pereira SN, Portela LOC, Cardoso DM, Lago PD, Dos Santos Guarda N, Moresco RN, Pereira MB, de Albuquerque IM. Moderate-to-high intensity inspiratory muscle training improves the effects of combined training on exercise capacity in patients after coronary artery bypass graft surgery: A randomized clinical trial. Int J Cardiol. 2019 Mar 15;279:40-46. doi: 10.1016/j.ijcard.2018.12.013. Epub 2018 Dec 10. PMID 30581100
- [Background] Miozzo AP, Stein C, Marcolino MZ, Sisto IR, Hauck M, Coronel CC, Plentz RDM. Effects of High-Intensity Inspiratory Muscle Training Associated with Aerobic Exercise in Patients Undergoing CABG: Randomized Clinical Trial. Braz J Cardiovasc Surg. 2018 Jul-Aug;33(4):376-383. doi: 10.21470/1678-9741-2018-0053. PMID 30184035
- [Background] Fernandez-Rubio H, Becerro-de-Bengoa-Vallejo R, Rodriguez-Sanz D, Calvo-Lobo C, Vicente-Campos D, Chicharro JL. Inspiratory Muscle Training in Patients with Heart Failure. J Clin Med. 2020 Jun 2;9(6):1710. doi: 10.3390/jcm9061710. PMID 32498445
- [Background] Sadek Z, Salami A, Joumaa WH, Awada C, Ahmaidi S, Ramadan W. Best mode of inspiratory muscle training in heart failure patients: a systematic review and meta-analysis. Eur J Prev Cardiol. 2018 Nov;25(16):1691-1701. doi: 10.1177/2047487318792315. Epub 2018 Aug 3. PMID 30073849
- [Background] Roncada G, Dendale P, Linsen L, Hendrikx M, Hansen D. Reduction in pulmonary function after CABG surgery is related to postoperative inflammation and hypercortisolemia. Int J Clin Exp Med. 2015 Jul 15;8(7):10938-46. eCollection 2015. PMID 26379888
- [Background] Haeffener MP, Ferreira GM, Barreto SS, Arena R, Dall'Ago P. Incentive spirometry with expiratory positive airway pressure reduces pulmonary complications, improves pulmonary function and 6-minute walk distance in patients undergoing coronary artery bypass graft surgery. Am Heart J. 2008 Nov;156(5):900.e1-900.e8. doi: 10.1016/j.ahj.2008.08.006. Epub 2008 Oct 5. PMID 19061704
- [Background] Cahalin LP, Arena RA. Breathing exercises and inspiratory muscle training in heart failure. Heart Fail Clin. 2015 Jan;11(1):149-72. doi: 10.1016/j.hfc.2014.09.002. PMID 25432483
- [Background] Kenji Nawa R, Daros Dos Santos T, Albiero Real A, Correa Matheus S, Tatsch Ximenes M, Machado Cardoso D, Martins de Albuquerque I. Relationship between Perme ICU Mobility Score and length of stay in patients after cardiac surgery. Colomb Med (Cali). 2022 Jul 30;53(3):e2005179. doi: 10.25100/cm.v53i3.5179. eCollection 2022 Jul-Sep. PMID 37152522
- [Background] Joseph P, Leong D, McKee M, Anand SS, Schwalm JD, Teo K, Mente A, Yusuf S. Reducing the Global Burden of Cardiovascular Disease, Part 1: The Epidemiology and Risk Factors. Circ Res. 2017 Sep 1;121(6):677-694. doi: 10.1161/CIRCRESAHA.117.308903. PMID 28860318
- [Background] Mummery RS, Rothschild M, Valadon LR. Carotenoids in two silk moths Saturnia pavonia L. and Actia luna L. Comp Biochem Physiol B. 1975 Jan 15;50(1):23-8. doi: 10.1016/0305-0491(75)90293-x. No abstract available. PMID 1122717

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 56 patients with CVD were screened. 32 declined to participate and 13 did not meet the inclusion criteria.
Period: Overall Study
Arm/Group | Study Group | Sham Group
Started | 5 | 6
Completed | 5 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Study Group | Sham Group | Total
Number analyzed (Participants) | 5 | 6 | 11
Age, Continuous [Mean (Standard Deviation); unit: Years] | 60.8 (9.9) | 60.5 (7.1) | 60.6 (8.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 2 | 4 | 6
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 36.1 (16.5) | 34.1 (5.9) | 35.0 (11.3)
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Inspiratory Muscle Function
Description: maximal inspiratory pressure (MIP) is the highest pressure measured during inspiration will be used.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: cm H2O
Arm/Group | Study Group | Sham Group
Number analyzed (Participants) | 5 | 6
cm H2O
  Baseline | 46.4 (13.4) | 52.8 (12.5)
  Post | 68.8 (13.6) | 50.0 (15.8)
Statistical Analysis 1: Comparison: Study Group vs Sham Group; Test type: Superiority; <0.001

2. Primary Outcome: Endothelial Function
Description: flow-mediated dilation (FMD) ultrasound measurements of brachial artery flow-mediated dilatation will be performed.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: Percentage
Arm/Group | Study Group | Sham Group
Number analyzed (Participants) | 5 | 6
Percentage
  Baseline | 5.41 (1.93) | 3.88 (2.26)
  Post | 7.53 (1.62) | 3.00 (1.51)
Statistical Analysis 1: Comparison: Study Group vs Sham Group; Test type: Superiority; p = .001, ANOVA

3. Primary Outcome: Arterial Stiffness
Description: arterial stiffness will be assessed by measuring pulse wave velocity.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: m per second
Arm/Group | Study Group | Sham Group
Number analyzed (Participants) | 5 | 6
m per second
  Baseline | 6.19 (0.53) | 5.57 (0.58)
  Post | 6.11 (0.56) | 5.58 (0.56)
Statistical Analysis 1: Comparison: Study Group vs Sham Group; Test type: Superiority; p = .001, ANOVA

4. Secondary Outcome: Functional Exercise Capacity
Description: maximal distance in 6 minute walk test will be used.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Study Group | Sham Group
Number analyzed (Participants) | 5 | 6
meters
  Baseline | 301 (39.8) | 309.2 (33.5)
  Post | 340.4 (36.6) | 305.0 (34.9)
Statistical Analysis 1: Comparison: Study Group vs Sham Group; Test type: Superiority; p < 0.001, ANOVA

5. Secondary Outcome: Dyspnea
Description: The modified Medical Research Council (mMRC) Dyspnea Scale, which have 5 points (0 to 4) will be used. High scores presented worsen dyspnea.
Time Frame: 4 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Study Group | Sham Group
Number analyzed (Participants) | 5 | 6
score
  Baseline | 2.8 (0.5) | 2.5 (0.6)
  Post | 1.6 (0.6) | 2.7 (0.5)
Statistical Analysis 1: Comparison: Study Group vs Sham Group; Test type: Superiority; p < 0.001, ANOVA

ADVERSE EVENTS:
Time Frame: From enrollment to the end of intervention
Arm/Group | Study Group | Sham Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/6
Other Adverse Events (participants affected / at risk) | 0/5 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT06127147/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-12): https://cdn.clinicaltrials.gov/large-docs/47/NCT06127147/SAP_003.pdf